CLINICAL TRIAL: NCT03295682
Title: Registry in Patients With Thoracoabdominal Aneurysms Treated With Multi-branch Stent Grafts Tailored to Their Individual Anatomies
Brief Title: Registry in Patients With Thoracoabdominal Aneurysms
Acronym: CONNECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CONNECT
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Thoracoabdominal Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular thoracoabdominal aneurysm repair — Endovascular treatment of patients with thoracoabdominal aneurysm using a multibranch stent graft tailored to the patient´s anatomy in combination with peripheral covered stents to bridge the visceral arteries

SUMMARY:
In this study patients will be observed, who receive a multi-branch stent graft tailored to the patients anatomy for the endovascular treatment of a thoracoabdominal aortic aneurysm Crawford type I, II, III, IV or V.

The objective of this study is to evaluate clinical and technical success as well as safety and feasibility of the multi-branch stent graft Systems used in endovascular treatment of thoracoabdominal aortic aneurysms that cannot be treated with commercially available devices. Primary endpoint of this study is the rate of patients with stable or decreasing aneurysm size at 12 months follow-up.

DETAILED DESCRIPTION:
In this study patients will be observed, who receive a multi-branch stent graft tailored to the patient´s anatomy for the endovascular treatment of a thoracoabdominal aortic aneurysm Crawford type I, II, III, IV or V. Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with a multi-branch stent graft produced by JOTEC GmbH. Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before data are being collected.

The period of data collection will be 36 months from the intervention for each patient. A risk based source data verification will be performed. CT angiograms will be evaluated by a CoreLab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients must have a thoracoabdominal aneurysm type Crawford type I, II, III, IV, or V
* Patients must have a suitable proximal landing area
* Patients must have a suitable distal landing area in the abdominal aorta or the iliac arteries
* Patients must have suitable access vessels
* Patients must be available for the appropriate follow-up times for the duration of the study
* Patients have signed the informed consent before intervention

Exclusion Criteria:

* Patients with infectious aneurysm
* Patients with inflammatory aneurysm
* Patients with ruptured or symptomatic aneurysm
* Patients with traumatic aneurysm
* Patients with aortic dissection
* Patients who have a congenital degenerative collagen disease or connective tissue disorder
* Patients with thrombocytopenia
* Patients with an eGFR < 45ml/min/1.73m2 before the intervention
* Patients with untreated hyperthyroidism
* Patients with malignancy needing chemotherapy or radiation
* Patients that will be treated or are treated with iliac branch devices
* Patients pre-treated with Nellix (Endologix) or Ovation (Endologix) or Altura (Lombard Medical) stent grafts
* Patients who are enrolled in another clinical study
* Patients with life expectancy of less than 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total number of 40 male and female patients with asymptomatic thoracoabdominal aortic aneurysm, treated with a multi-branch stent graft system.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with stable or decreasing aneurysm size at 12 months follow-up (measured by CoreLab) | 12 months follow-up
  Decreasing size: >/= 5mm Increasing size: </= 5mm compared to first post-operative CT angiogram

SECONDARY OUTCOMES:
Rate of all cause mortality | intra-op, post-op until 36 months follow-up
Rate of patients with aneurysm rupture | post-op until 36 months follow-up
Rate of patients with main adverse events (product-related, procedure-related, aneurysm-related) | post-op until 36 months follow-up
Rate of interventions in peri-operative periods (all related interventions until index procedure) | intra-op
Rate of reinterventions | post-op until 36 months follow-up
Rate of patients with endoleaks type Ia, Ib, II, III, IV, V and of unknown origin | post-op until 36 months follow-up
Rate of patients with multi-branch stent graft migration | post-op until 36 months follow-up
Rate of patients with loss of device integrity | post-op until 36 months follow-up
Rate of patients with primary / secondary patency of branch vessels | post-op until 36 months follow-up
Rate of patients with stent graft infection | post-op until 36 months follow-up
Rate of patients with primary / secondary technical success | post-op until 36 months follow-up
Rate of patients with primary / secondary clinical success | post-op until 36 months follow-up
Rate of patients with removal or failure to implant the multi-branch stent graft | intra-op, post-op until 36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Schelzig, Professor, Study Director — Uniklinikum Düsseldorf
Locations (1):
- Uniklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany